CLINICAL TRIAL: NCT03637816
Title: Qualitative Study on Experiences Related to Anorexia and the Effects of Anamorelin and Placebo in Advanced Non-Small-Cell Lung Cancer Patients With Anorexia-Cachexia: A Preliminary Study
Brief Title: Anamorelin Hydrochloride in Reducing Anorexia in Patients With Advanced Non-small Cell Lung Cancer
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2017-1059; NCI-2018-01593 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2017-1059 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2018-08-10; First posted 2018-08-20 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Anorexia; Lung Non-Small Cell Carcinoma; Stage III Lung Cancer AJCC v8; Stage IIIA Lung Cancer AJCC v8; Stage IIIB Lung Cancer AJCC v8; Stage IIIC Lung Cancer AJCC v8; Stage IV Lung Cancer AJCC v8; Stage IVA Lung Cancer AJCC v8; Stage IVB Lung Cancer AJCC v8
MeSH Terms: conditions — Anorexia; Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — anamorelin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (anamorelin hydrochloride) (Experimental): Patients receive anamorelin hydrochloride PO daily for 9 weeks in the absence of disease progression or unaccepted toxicity.
  Interventions: Drug: Anamorelin Hydrochloride; Other: Questionnaire Administration
- Arm II (placebo) (Placebo Comparator): Patients receive placebo PO daily for 9 weeks in the absence of disease progression or unaccepted toxicity.
  Interventions: Other: Placebo; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Anamorelin Hydrochloride — Given PO
  Other Names: RC-1291 HCl
  Arms: Arm I (anamorelin hydrochloride)
Other: Placebo — Given PO
  Other Names: placebo therapy; PLCB; sham therapy
  Arms: Arm II (placebo)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II/III trial studies how well anamorelin hydrochloride works in reducing anorexia in patients with non-small cell lung cancer that has spread to other places in the body. Anamorelin hydrochloride may help to improve patients' appetite in order to stop weight loss.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To qualitatively examine experiences related to anorexia in advanced lung cancer patients with anorexia-cachexia and the impact of nine weeks of treatment of oral anamorelin hydrochloride (anamorelin) (100 mg) and placebo.

SECONDARY OBJECTIVES:

I. To explore changes in anorexia-cachexia (measured by the Functional Assessment of Anorexia/Cachexia Treatment [FAACT] anorexia/cachexia subscale [A/CS]) in patients with advanced non-small cell cancer after 9 weeks of oral anamorelin (100 mg) or placebo.

II. To explore changes in anorexia as measured by the 5-item Anorexia Symptom score (derived from the FAACT A/CS) after 9 weeks of oral anamorelin (100 mg) or placebo.

III. To explore any associations between changes in anorexia with body weight, body composition (as assessed by InBody, weight scale, and L3 vertebrae compute tomography [CT] scan), quality of life (Functional Assessment of Cancer Illness Therapy [FACT-G]), Patient Global Impression of Severity (PGIS), Patient Global Impression of Change (PGIC), nutritional markers (pre-albumin, IGF-1 and IGFBP-3), inflammatory biomarkers (C-reactive protein [CRP], monocyte IL-6&R, TNF-a&R, IL-10,IL-8, IL-1&RA), and food intake after 9 weeks of oral anamorelin (100 mg) or placebo.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive anamorelin hydrochloride orally (PO) daily for 9 weeks in the absence of disease progression or unaccepted toxicity.

ARM II: Patients receive placebo PO daily for 9 weeks in the absence of disease progression or unaccepted toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of advanced non-small cell lung cancer
* Presence of anorexia, defined as =< 37 points on FAACT A/CS domain (on a 0 to 48-point scale in which 0 = worst possible anorexia/cachexia)
* Patients with a history of either: >= 5% of weight loss for body mass index (BMI) >= 20 kg/m^2 or >= 2% of weight loss for BMI < 20 kg/m^2, over a period of 1 year
* Patients must be willing to keep a daily medication diary and engage in telephone follow up with research staff
* Patients must have telephone access to allow contact by the research staff
* Adequate hepatic function, defined as aspartate transaminase (AST) and alanine transaminase (ALT) levels =< 5 x upper limit of normal (ULN)
* Life expectancy of >= 6 months

Exclusion Criteria:

* Major contraindication to anamorelin i.e. hypersensitivity
* BMI >= 28 kg/m^2
* Inability to complete the baseline assessment forms or to understand the recommendations for participation in the study
* Pregnant or lactating women. Women of childbearing age not on birth control. For inclusion in the study, a negative pregnancy test for women of childbearing potential, as defined by intact uterus and at least one ovary, and a history of menses within the last 12 months is necessary. Pregnancy test is to be performed no greater than 14 days prior to consent in study. In cases of women with elevated b-human chorionic gonadotropin (HCG), these candidates will be eligible to participate so long as the level of b-HCG is not consistent with pregnancy. Women of childbearing potential must be on or use contraception during the study period. Their male partners must also use contraception (condom) or maintain abstinence. Birth control specifications: Women who are able to become pregnant must use birth control during the study and for 30 days after the last anamorelin dose. Acceptable forms of birth control include barrier methods (such as condom or diaphragm) with spermicide
* Uncontrolled diabetes mellitus (fasting blood sugar > 200 mg/dl) at screening
* Patients on drugs with strong CYP 3A4 inhibitors within the previous two weeks (ketoconazole, clarithromycin, itraconazole, nefazodone, telithromycin)
* Patients on drugs that may prolong the PR or QRS interval durations, such as any of the class I/sodium (Na+) channel blocking antiarrhythmic medications should be avoided (e.g. flecainide, procainamide, propafenone, quinidine)
* Patients currently on investigational therapies will be evaluated by the principal investigator (PI) on a case by case basis and study participation approval will be obtained from the treating oncologist
* Patient currently taking androgenic compounds (including but not limited to testosterone, testosterone-like agents, oxandrolone, megestrol acetate, methylphenidate, corticosteroids [note: topical, inhaled, or oral corticosteroids taken for a short duration (=< 5 consecutive days) after chemotherapy are acceptable]), dronabinol or medical marijuana (medical cannabis) or any other prescription medication or off-label products intended to increase appetite or treat unintentional weight loss
* Any relevant condition that would interfere with ability to participate in one-on-one interviews either in person or via telephone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-11-27 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
To reach thematic saturation by qualitatively examining experiences related to anorexia at the baseline in advanced lung cancer patients with anorexia/cachexia receiving either oral Anamorelin 100 mg or placebo. | Baseline up to day 64
  A 60-90 minute interview will be conducted to identify and explore a range of issues, including: impact on daily psycho-social function (relationships, work, mood, initiative, pleasurable activities); food intake; independence; physiological changes in appetite/eating; visuality of cachexia; weight loss interpreted as a "bad sign"; response from health care professionals; conflict over food; coping responses; and the patient's report of meaningful change in symptoms due to the intervention (and if so, why).

SECONDARY OUTCOMES:
Explore changes in anorexia/cachexia in patients with advanced non-small cell cancer after oral anamorelin 100 mg/placebo treatment | Baseline up to day 64
  Measured by the Functional Assessment of Anorexia/Cachexia Treatment (FAACT) anorexia/cachexia subscale (A/CS). The FAACT A/CS domain is a 12-item symptom-specific domain designed to measure patients' additional concerns about their anorexia /cachexia during the previous 7 days on a scale of 0 to 4.
Explore changes in anorexia after 9 weeks of oral Anamorelin 100 mg or placebo treatment | Baseline up to day 64
  Measured by the A/CS. 5-item Anorexia Symptom Scale obtained by summing 5 anorexia symptom items derived from the FAACT A/CS domain measured by the following responses: "good appetite," "interest in food drops," "food tastes unpleasant," "get full quickly," and "difficulty eating rich/heavy foods".
Explore associations between changes in anorexia and body composition assessed with body weight in kilograms and (lean body mass in kilograms). | Baseline up to day 64
  Body weight and height will be combined to report BMI in kg/m^2
Explore associations between changes in anorexia with nutrition assessed by serum pre-albumin, Insulin Growth Factor-1 (IGF-1), and IGF binding protein-3 (IGFBP-3). | Baseline up to day 64
  Measured by blood proteins to evaluate nutrition improvement related to loss of appetite and body weight loss.
Explore associations between changes in anorexia with inflammation assessed by C-Reactive Protein (CRP), monocyte IL-6&R, TNF-α&R, IL-10,IL-8,IL-1&RA) inflammatory biomarkers. | Baseline up to day 64
  Measured by blood proteins (cytokines) to evaluate inflammation improvement related to loss of appetite and body weight loss.
Explore associations between changes in anorexia with quality of life assessed by Functional Assessment of Cancer Illness Therapy (FACT-G) | Baseline up to day 64
  The FACT-G is a 27-item compilation of general questions divided into four primary domains: Physical Well-Being, Social/Family Well-Being, Emotional Well-Being, and Functional Well-Being. Answers rated from 0 meaning "Not at All" to 4 meaning "Very Much".
Explore any associations between changes in anorexia assessed by Patient Global Impression of Severity (PGIS) Scale | Baseline up to day 64
  PGIS is a validated global impression scales used to evaluate subjective patients' response at the end of the intervention by assessing the severity and change in the symptom of interest. Determined by the participant's responses: Which of the following statements best describes your current appetite/eating-related symptoms? I currently do not have any appetite/eating-related symptoms I currently have minor appetite/eating-related symptoms I currently have moderate appetite/eating-related symptoms I currently have severe appetite/eating-related symptoms..
Explore any associations between changes in anorexia assessed by Patient Global Impression of Change (PGIC) | Baseline up to day 64
  PGIC is a validated global PGIC is a validated global impression scales used to evaluate subjective patients' response at the end of the intervention by assessing the severity and change in the symptom of interest using the following questions: "Since the start of the treatment, how would you describe your change in appetite/eating-related symptoms?" and "Since the start of treatment, how would you describe your change in your overall condition?" Determined by participant's responses ranging from "Very Much Improved" to "Very Much Worse".
Explore any associations between changes in anorexia with food intake after 9 weeks of oral Anamorelin 100 mg or placebo treatment | Baseline up to day 64
  Participants will record their food and beverage intake at the time of consumption using MyFitnessPal.

CONTACTS AND LOCATIONS:
Overall Officials: Sriram Yennu, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Yennurajalingam S, Mott F, Lu Z, Urbauer D, Stanton P, Torres H, Rantanen PA, Davis S, Dev R, Hui D, Bruera E. Perception of subjective lived experiences of individuals with anorexia-cachexia in patients with advanced lung cancer. Asia Pac J Oncol Nurs. 2023 Oct 10;10(Suppl 1):100314. doi: 10.1016/j.apjon.2023.100314. eCollection 2023 Nov. PMID 38197040
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org